CLINICAL TRIAL: NCT07367685
Title: Clinical Study of Universal CD19 CAR-γδT Cell Injection in the Treatment of Adult Relapsed/Refractory B-cell Lymphoma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Second Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Meiling Li, The Chief of the Department of Hematology, The Second Affiliated Hospital of Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QH10309-NHB-01（0）
Record Dates: First submitted 2026-01-05; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Recurrent/Refractory B-cell Lymphoma
Keywords: CD19; CAR-γδT; cell therapy
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult patients with relapsed/refractory CD19-positive B-cell lymphoma (Experimental): A conditional chemotherapy regimen of fludarabine and cyclophosphamide will be administered, followed by investigational therapy, QH103 Cells
  Interventions:
  Biological: QH103 Cell Injection Drug: Fludarabine Drug: Cyclophosphamide
  Interventions: Biological: QH103 Cell Injection; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: QH103 Cell Injection — Biological: CD 19-CAR T cell Following lymphodepletion with chemotherapy (cyclophosphamide and fludarabine) patients will be treated with dose escalation (3+3) : dose 1 (3×10^8 CAR+cells) ,dose 2 (6× 10^8 CAR+cells).
  Other Names: CD19CAR-γδT cell injection
Drug: Cyclophosphamide — Eligible subjects will undergo lymphodepletion chemotherapy 5 to 3 days prior to cell infusion. The recommended lymphodepletion regimen comprises cyclophosphamide (500-1000 mg/m² administered 3 days).
Drug: Fludarabine — Eligible subjects will receive lymphodepletion chemotherapy 5 to 3 days prior to cell infusion. The recommended lymphodepletion regimen comprises fludarabine (30-40 mg/m² administered 3 days).

SUMMARY:
This study is an open-label, single-arm clinical trial designed to evaluate the safety and tolerability of QH103 cell injection solution in adult subjects with relapsed/refractory CD19-positive B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, no gender restrictions;
* Clinically diagnosed with relapsed/refractory B-cell lymphoma, malignant B- cell lymphoma (according to the Lugano (2014) criteria, with at least one evaluable tumour lesion, defined as: Lymph node lesions with a longest diameter exceeding 1.5 cm, or extranodal lesions with a longest diameter exceeding 1.0 cm), including diffuse large B-cell lymphoma (DLBCL-NOS), encompassing activated B-cell (ABC)/grossly centre B-cell (GCB) subtypes, primary mediastinal (thymic) large B-cell lymphoma (PMBCL), transformative follicular lymphoma (TFL), high-grade B-cell lymphoma (HGBCL) with MYC and BCL2 and/or BCL6 rearrangements,follicular lymphoma (FL), mantle cell lymphoma (MCL), marginal zone lymphoma (MZL)

  1. Relapsed B-cell lymphoma is defined as disease progression following ≥2 systemic therapies;
  2. Refractory disease is defined as failure to achieve complete remission (CR) on first-line therapy, or best response to first-line therapy being disease progression (PD), or best response after at least 4 cycles of first-line therapy being stable disease (SD)(e.g., 4 cycles of R-CHOP), or best response after at least 6 cycles being partial remission (PR) with biopsy-confirmed residual disease or disease progression within ≤6 months of treatment.
* Cytologically or histologically confirmed CD19-positive tumour cell immunophenotyping;
* Expected survival exceeding 3 months;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
* Major organ function meeting the following criteria: Echocardiogram showing left ventricular ejection fraction ≥50%; serum creatinine ≤ 1.5 × upper limit of normal (ULN); alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ 3 × ULN; total bilirubin ≤ 1.5 × ULN;
* Negative pregnancy test for women of childbearing potential; both male and female subjects must agree to use effective contraception during treatment and for 1 year thereafter;
* Toxicity from prior antineoplastic therapy ≤ Grade 1 (per CTCAE version 5.0) or acceptable to the inclusion/exclusion criteria;
* No significant hereditary disorders;
* Ability to comprehend trial requirements and procedures, with willingness to participate in the clinical study as directed;
* Signing of the trial informed consent form.

Exclusion Criteria：

* Presence of central nervous system (CNS) involvement or clinically significant history of CNS disorders, such as epilepsy and cerebrovascular disease;
* Pregnant or lactating women, or women unwilling to use effective contraception during treatment and for 1 year post-treatment;
* Unremitted other malignancies;
* Patients with primary immunodeficiency or autoimmune diseases requiring immunosuppressive therapy;
* Patients who received allogeneic immune cell therapy within 6 months prior to enrolment, or donor lymphocyte infusion within 6 weeks prior to enrolment;
* Confirmed serum reactivity positive for anti-FMC63 and DSA;
* Patients participating in other clinical trials within 4 weeks prior to enrolment;
* Uncontrolled infectious diseases or other serious conditions, including but not limited to infections (Human Immunodeficiency Virus, acute or chronic active hepatitis B or C), congestive heart failure, unstable angina pectoris, arrhythmias, or conditions deemed to pose unpredictable risks by the treating physician;
* History of stroke or intracranial haemorrhage within 3 months prior to enrolment;
* Major surgery or trauma within 28 days prior to enrolment, or unresolved significant adverse events;
* History of allergy to any component of the cell product;
* Inability to comprehend or unwillingness to sign the informed consent form;
* Other reasons deemed by the investigator to render the patient unsuitable for the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Event | 12months
  AE is defined as any adverse medical event from the date of leukapheresis to 12 months after QH103 infusion. Among them, cytokine release syndrome (CRS) and immune cell-associated neurotoxicity syndrome (ICANS) were graded according to American Society for Transplantation and Cellular Therapy (ASTCT) criteria, graft-versushost disease (GVHD) according to criteria defined by the Mount Sinai Acute GVHD International Consortium. Other AEs were graded according to common terminology criteria for adverse events (CTCAE) v5.0
Incidence of Dose-Limiting Toxicities (DLTs) | First infusion date of QH103 cells to 28 days end cell infusion
  DLT was defined as QH103 Cells-related events with onset within first 28 days following infusion.
Maximum tolerated dose (MTD) | 28 days
  MTD is defined as the highest dose level of less than or equal to 2 DLT among the 6 subjects finally determined.

SECONDARY OUTCOMES:
PK-Tmax | 12 months
  Time to peak in CAR-T cell count in peripheral blood after infusion of QH103.
Pharmacodynamics: Peak level of cytokines in serum | 12 months
  The Changes from baseline of level cytokines and chemokines in peripheral blood after infusion of QH103
Overall Response Rate(ORR) | 6 months
  Defined as complete response plus partial response.
Overall Survival（OS） | 6 months&12 months
  Survival as estimated by Kaplan-Meier method. Death from any cause is considered as event for analysis.
Progression-Free Survival（PFS） | 6 months
  Survival as estimated by Kaplan-Meier method. The length of time during and after the treatment of a disease is considered as event for analysis.
PK-Cmax | 12 months
  Peak concentration (Cmax) in the CAR-T cell count in peripheral blood after infusion of QH103.
PK-AUC | 12 months
  Area under the concentration-time curve of CAR-T cell count in peripheral blood after infusion of QH103 from 0 to 12 months
PK-Tlast | 12 months
  The final time point in CAR-T cell count in peripheral blood after infusion of QH103.
PK-Clast | 12 months
  The final point concentration (C last) in the CAR-T cell count in peripheral blood after infusion of QH103

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Fujian Medical University, Quanzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided
If used for publication in academic papers, data that does not involve the personal privacy of research subjects will be provided in accordance with journal requirements.